CLINICAL TRIAL: NCT06765330
Title: Microbiome Changes Following Laser and Chlorhexidine Cavity Disinfection in Different Caries Removal Methods
Brief Title: Microbiome Changes After Laser and Chlorhexidine Disinfection in Caries Removal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ayse Tugba Erturk Avunduk, Associate Profesor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MersinU-DHF-ATEA-01
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries
Keywords: dental caries; disinfection; laser; chlorhexidine gluconate; pyrosequencing
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Group 1: Non-selective caries removal with tungsten carbide bur + No cavity disinfection Group 2: Non-selective caries removal with tungsten carbide bur + 2% chlorhexidine disinfection Group 3: Non-selective caries removal with tungsten carbide bur + Er, Cr: YSGG laser disinfection Group 4: Selective caries removal with polymer bur + No cavity disinfection Group 5: Selective caries removal with polymer bur + 2% chlorhexidine disinfection Group 6: Selective caries removal with polymer bur + Er, Cr: YSGG laser disinfection
Who Masked: Participant
Masking Description: The randomization of the participants for this study will be carried out on the previously determined date and time using the address https://randomizer.org/
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: Non-selective caries removal with tungsten carbide bur + No cavity disinfection (Active Comparator): Access to the lesion will be achieved using a high-speed handpiece with a sterile high-speed bur (#245 bur Meisinger GmbH, Germany). The caries removal strategy towards soft dentin will be performed following the guidelines published by the International Caries Consensus Collaboration. The caries will be completely removed from the surrounding cavity walls with a tungsten carbide bur, leaving at least 2 mm of peripheral intact tooth structure for good adaptation and sealing of the restoration. Superficial necrotic caries fragments, which deform when an instrument is pressed into them and can be easily removed with little force, will be removed from the pulpal floor using a sharp sterile excavator, while soft dentin will be left at the cavity floor to avoid pulpal exposure.
  Following caries removal, the tooth will be restored without any cavity disinfection.
  Interventions: Procedure: Tungsten carbide bur
- Group 2: Non-selective caries removal with tungsten carbide bur + 2% chlorhexidine disinfection (Active Comparator): Following the caries removal protocol applied in Group 1, 2% chlorhexidine (Consepsis®, Ultradent) will be applied to the cavity for 20 seconds. The cavity will then be air-dried for 10 seconds, and the tooth will be restored.
  Interventions: Drug: CHX disinfection; Procedure: Tungsten carbide bur
- Group 3: Non-selective caries removal with tungsten carbide bur + Er,Cr: YSGG laser disinfection (Active Comparator): Following the caries removal protocol applied in Group 1, the cavity will be disinfected using an Er,Cr: YSGG laser (EPIC X™, BIOLASE, USA) with 940 nm and 0.1 W output power. Then, the tooth will be restored.
  Interventions: Device: Laser Disinfection; Procedure: Tungsten carbide bur
- Group 4: Selective caries removal with polymer bur + No cavity disinfection (Active Comparator): Access to the lesion will be achieved using a high-speed handpiece with a sterile high-speed bur (#245 bur Meisinger GmbH, Germany). The SS White Smartburs II® will be used with a low-speed handpiece at 5,000-10,000 RPM to remove carious dentin of sizes RA4, RA6, and RA8 depending on the size of the caries lesion. The instrument will be used with a circular, light force starting from the center of the carious lesion towards the periphery as recommended by the manufacturer. Caries removal will be stopped when the instrument is macroscopically worn and blunt and can no longer remove tissue. An explorator will be used to verify if any caries remain at the base of the cavity. If necessary, a new polymer bur, SmartbursII®, will be used to remove the remaining decay.
  After selective caries removal, the tooth will be restored without any cavity disinfection.
  Interventions: Procedure: Polymer bur
- Group 5: Selective caries removal with polymer bur + 2% chlorhexidine disinfection (Active Comparator): Following the selective caries removal protocol applied in Group 4, 2% chlorhexidine (Consepsis®, Ultradent) will be applied to the cavity for 20 seconds. The cavity will then be air-dried for 10 seconds, and the tooth will be restored.
  Interventions: Drug: CHX disinfection; Procedure: Polymer bur
- Group 6: Selective caries removal with polymer bur + Er,Cr: YSGG laser disinfection (Active Comparator): Following the selective caries removal protocol applied in Group 4, the cavity will be disinfected using an Er, Cr: YSGG laser (EPIC X™, BIOLASE, USA) with 940 nm and 0.1 W output power. Then, the tooth will be restored.
  Interventions: Device: Laser Disinfection; Procedure: Polymer bur

INTERVENTIONS:
Drug: CHX disinfection — Each CHX cavity will be treated with disinfectant with a disposable micro brush tip and left undisturbed for 20 seconds. They will then be air-dried for 10 seconds and restore the tooth.
  Arms: Group 2: Non-selective caries removal with tungsten carbide bur + 2% chlorhexidine disinfection; Group 5: Selective caries removal with polymer bur + 2% chlorhexidine disinfection
Device: Laser Disinfection — After the caries removal procedure, the cavity will be disinfected using an Er,Cr: YSGG laser (EPIC X™, BIOLASE, USA) with 940 nm and 0.1 W output power. The laser tip will be a 400 µm tip with an energy density of 138.12 J/cm in non-contact mode (2 mm distance), 5 s/mm2 sweeping motion.
  Arms: Group 3: Non-selective caries removal with tungsten carbide bur + Er,Cr: YSGG laser disinfection; Group 6: Selective caries removal with polymer bur + Er,Cr: YSGG laser disinfection
Procedure: Tungsten carbide bur — Carious tissue will be completely removed from the surrounding cavity walls with a tungsten carbide bur, leaving at least 2 mm of peripheral intact tooth structure for good adaptation and sealing of the restoration.
  Arms: Group 1: Non-selective caries removal with tungsten carbide bur + No cavity disinfection; Group 2: Non-selective caries removal with tungsten carbide bur + 2% chlorhexidine disinfection; Group 3: Non-selective caries removal with tungsten carbide bur + Er,Cr: YSGG laser disinfection
Procedure: Polymer bur — Access to the lesion will be achieved using a high-speed handpiece with a sterile high-speed bur. The polymer bur will be used with a low-speed handpiece at 5,000-10,000 RPM to remove carious dentin in sizes RA4, RA6, and RA8 according to the size of the caries lesion. The instrument will be used with a circular, light force starting from the center of the carious lesion towards the periphery as recommended by the manufacturer. Caries removal will be stopped when the instrument is macroscopically worn and blunt and can no longer remove tissue. An excavator will be used to verify if any caries remain at the base of the cavity. If necessary, a new polymer bur will be used to remove the remaining decay.
  Arms: Group 4: Selective caries removal with polymer bur + No cavity disinfection; Group 5: Selective caries removal with polymer bur + 2% chlorhexidine disinfection; Group 6: Selective caries removal with polymer bur + Er,Cr: YSGG laser disinfection

SUMMARY:
The aim of this study was to investigate the effects of cavity disinfection with laser and chlorhexidine on the microbiome in cavities prepared using different caries removal methods.

DETAILED DESCRIPTION:
Prevention and treatment of dental caries, one of the most common and oldest diseases, is closely related to human health. Dental hard tissue undergoes remineralization and demineralization processes in a cycle. Caries occur when this balance is disturbed in favor of demineralization. Dental caries is the loss of minerals caused by the acid produced by microorganisms.

In conventional caries removal, high-speed rotating hand instruments are generally used to reach the lesion. In contrast, low-speed rotating hand instruments (tungsten carbide burs) remove the caries. This method involves rapid and efficient caries removal but may result in the removal of healthy tissue or affected dentin capable of remineralization. During minimally invasive procedures, more sparing and selective methods of caries removal are widely used in operative dentistry as an alternative to the conventional method. One of these methods is polymer burs produced as an alternative to conventional tungsten carbide burs. They are made of soft polymer material. It removes only infected dentin. Polymer burs are harder than carious dentin and softer than healthy dentin. Therefore, when removing carious tissue with a polymer bur, the bur remains intact, but when it comes to healthy tissue, the bur wears out. It is designed to remove only carious dentin by selectively maintaining its cutting efficiency until it encounters caries-affected dentin. In a previous study, microbiological Streptococcus mutans bacteria count reduction before and after occlusal caries removal was statistically significant with polymer burs compared to tungsten carbide burs.

In restorative dentistry, complete removal of infected caries tissue before the restoration process plays a key role in the success of the treatment. Due to the risk of removing healthy dentin tissue while removing infected caries tissue, protective cavity preparation techniques have been developed. Criteria such as color and hardness, which are considered in the decision to remove caries from dental tissue, are subjective and depend on the senses of sight and touch. Although researchers recommend the use of caries indicators based on objective data, studies have shown that indicators are only 15-40% successful in detecting the presence of microorganisms. Despite the removal of the stained tissues, the presence of microorganisms was observed in the area close to the pulp, especially in the dentinal tubules. These microorganisms remaining in the tissue may cause secondary caries formation, postoperative sensitivity, and pulpal inflammation. Studies have shown that the occlusive and sealing properties of the restoration material cannot prevent the residual bacteria in the smear layer and dentinal canals from diffusing into the pulp tissue and causing infection. Therefore, the use of antibacterial cavity disinfectants has come to the fore. Today, chlorhexidine digluconate (CHX), benzalkonium chloride, sodium hypochlorite, hydrogen peroxide, iodine solutions, phosphoric acid, fluoride, propolis, ozone, light-activated disinfection systems, and laser systems are used as cavity disinfectants.

The microbiology of dental caries is a subject that has been studied for many years. Previous studies have used traditional culture-based methods to identify bacteria associated with dental caries. The culture-based method has allowed a basic understanding of the composition of dental plaque microbiota in dental caries. Microorganisms have been isolated from carious lesions or dental plaque samples collected from a cross-sectional or longitudinal study using culture-based techniques. However, research on the oral microbiome is still incomplete as artificial media cannot fully mimic the natural environment in which oral bacteria are found, because about half of the oral microbiome cannot be cultured. Therefore, it is not possible to detect all bacteria in the sample in studies using the culture method. Molecular genetic techniques can detect and identify the microbiome without culture using the analysis of 16s rRNA found in all these prokaryotes. The 16s rRNA gene is used as a standard for the classification and identification of the microbiome because 16s rRNA gene sequences contain hypervariable regions that can provide species-specific sequences for the identification of bacteria. Although initially used to identify bacteria, 16s rRNA sequencing was later used to reclassify bacteria into new species or genera. It has also been used to identify new species that have not yet been successfully cultured. Recently, high-throughput pyrosequencing has revealed unexpectedly high diversity within the human oral microbiome. Molecular genetic techniques have been used to detect and identify microorganisms in permanent teeth, necrotic pulp and periapical lesions, and clinical samples without direct culture.

The understanding of caries microbiology has been greatly enriched in recent years by the advancement of sequencing-based technology and bioinformatic analysis. However, there are no studies in the literature evaluating microbiome analysis in combination with different caries removal techniques and cavity disinfection methods. Therefore, this study aims to review the classical concepts of microbiological aspects of dental caries and to investigate the effects of cavity disinfection with laser and chlorhexidine on the microbiome in cavities prepared using different caries removal methods.

ELIGIBILITY:
Inclusion criteria:

* Permanent molar/premolar teeth in which the carious lesion is on the occlusal surface and extends to the middle third of the dentin at most
* Individuals with good oral hygiene
* Absence of clinical symptoms of periapical pathology
* Teeth in occlusion with the opposite tooth
* Individuals born in 2007 and before (>18 years)
* Those who signed the Informed Voluntary Consent Form/Written Consent Form

Exclusion criteria:

* Irregular attendance at dental check-ups
* Severe systemic disease, allergy, and saliva flow disorder
* Poor oral hygiene
* Advanced periodontal disease
* Presence of clinically detected pulpal/periapical pathology
* Devitalisation of teeth
* The individual was born after 2007 (<18 years)
* Those who do not sign the Informed Voluntary Consent Form/Written Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Microbiome Changes | 3 months
  In all groups, dentin samples will be taken from the affected dentin at the base of the cavity as a result of three different subgroup disinfection procedures applied after the caries removal method using 2 sterile number 6 round sterile steel roun burs moistened with saline for microbial analysis. The burs will be placed in 5 ml sterile vials and stored at -80 0C until the analyses are performed. The prepared cavities will be completed with routine and standard treatment protocols. Following the finishing and polishing procedures, occlusion will be checked. The samples collected during the research process will be delivered to the A&D Genetic Diseases Evaluation Centre (Ankara, Turkey) where DNA isolation and sequence analysis will be performed together with molecular biologists. In the method, following the extraction of total genomic DNA from clinical samples, broad-range 16S rRNA PCR will be performed and MicroSeq 500 16S rRNA Sequencing kit will be used for sequence analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Tugba Erturk Avunduk, Associate Profesor, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Faculty of Dentistry, Department of Restorative Dentistry, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No